CLINICAL TRIAL: NCT05565547
Title: Clinical Validation Study for Multimodal Equipment for Teleophthalmology Assessment (META) Device
Brief Title: Multimodal Equipment for Teleophthalmology Assessment (META)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: IIT2022123
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Eye Diseases
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with common eye diseases: Patients who have common eye diseases, including common anterior segment eye diseases (conjunctivitis, keratitis, corneal opacity, cataract) and fundus diseases (age-related macular degeneration, diabetic retinopathy) and refractive error (myopia, high myopia, hyperopia, anisometropia and presbyopia).
  Interventions: Device: META; Device: Commercial devices

INTERVENTIONS:
Device: META — The META device is used for a comprehensive ophthalmic examination.
Device: Commercial devices — Commercial devices (including near and far eye charts, refractometer, optical biometry, slit lamp microscopy, fundus camera and OCT) are used for a comprehensive ophthalmic examination.

SUMMARY:
We have developed a Multimodal Equipment for Teleophthalmology Assessment (META) device. This novel device is compact, portable and suitable for packaging and express delivery. With this device, there is a potential to implement a new concept of "hospital-at-home" eye care model. The present study is designed to validate the META device for future clinical usage and investigation. We will compare the performance of the META device with those provided by commercial devices in terms of image quality of optical coherence tomography (OCT), anterior segment and fundus camera, and evaluate the level of agreement in lesion detection and quantitative measurements between META and other commercial devices (e.g., Heidelberg Spectralis OCT, Haag-Streit BQ900 Slit-lamp imaging, Canon CR-2 fundus imaging, Zeiss IOL Master 500).

DETAILED DESCRIPTION:
The META is an innovative and non-invasive examination instrument for a variety of common eye diseases. The integrated multimodality device combines digital slit lamp, fundus camera, OCT, refractometer, optical biometry and visual acuity test (near and distance) that facilitate a comprehensive ophthalmic examination. In the current study, all participants will undergo the measurements provided by the META and by traditional examination modalities (including digital slit lamp, fundus camera, OCT, refractometer, optical biometry and visual acuity test) in a random order. The participants will need to complete several questionnaires to investigate their preference and confidence to receive the META exams in the future.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older.
* Participants with healthy eyes, or patients diagnosed with one or more common eye diseases, including anterior segment eye diseases (conjunctivitis, keratitis, corneal opacity or cataract), fundus diseases (age-related macular degeneration or diabetic retinopathy) and/or refractive error (myopia, high myopia, hyperopia, anisometropia, or presbyopia).
* Willing and able to participate in all examinations related to this study
* Visual acuity of 20/400 or better in the study eye(s).

Exclusion Criteria:

* Ocular trauma or postoperative eyes within 3 months.
* Study eye(s) with dilated pupil.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with healthy eyes or with common eye diseases.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2022-10-15 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
Image Quality | in the same 1 day
  To evaluate the image quality of the META versus commercial devices. These images include slit-lamp anterior-segment images, colour fundus photographs, and OCT scans. The image quality metrics (e.g., position, focus, contrast, etc.) will be identified by masked qualified ophthalmologists independently and scored according to the same grading scheme
Level of agreement in quantitative measurements provided by META-OCT and by commercial OCT | in the same 1 day
  OCT images will be captured by META-OCT and by a commercial OCT, and segmented and analyzed with default algorithm to yield quantitative measurements.

SECONDARY OUTCOMES:
Level of agreement in axial length measurement | in the same 1 day
  Accuracy of axial length measurement will be captured by META-AL versus by a commercial biometric device.
Level of agreement in spherical equivalent diopter (SED) and astigmatism vector components (J0 and J45) | in the same 1 day
  Accuracy of SED and J0 and J45 will be obtained by META-SE versus by a commercial refractor.
Level of agreement in near and far visual acuity measurements | in the same 1 day
  Accuracy of near and far visual acuity measurements will be obtained by META-VA versus by reference ETDRS charts.
Level of agreement in detecting ocular abnormalities. | in the same 1 day
  Agreement in the detection of ocular abnormalities (e.g., corneal scars, keratic precipitates, lens opacification, macular fluid, or other retinopathy) by META images versus by commercial imaging devices.
Repeatability in quantitative measurements provided by META-OCT | in the same 1 day
  OCT images will be captured by META-OCT twice, and the repeatability of quantitative measurements will be assessed.
Exam success rate | in the same 1 day
  The exam success rate will be obtained by META versus by commercial devices.
Time spent on the examinations | in the same 1 day
  The time spent on the examinations will be obtained by META versus by commercial devices.
Patient experience | in the same 1 day
  Investigator-administered questionnaires will be used to investigate participants' preferences and confidence to receive META exams in the future.

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, M.D., Ph.D., Study Chair — State Key Laboratory of Ophthalmology, Zhongshan Ophthalmic Center, Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No